CLINICAL TRIAL: NCT03611283
Title: Topical Products to Treat Xerostomia in Primary Sjögren's Syndrome: a Double-blind Clinical Trial
Brief Title: Topical Management of Xerostomia With Dry Mouth Products
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rosa María López-Pintor Muñoz (Other)
Responsible Party: Sponsor-Investigator, Rosa María López-Pintor Muñoz, Associate Professor; Co-director Speciality in Oral Medicine, Universidad Complutense de Madrid
Organization: Universidad Complutense de Madrid (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0001
Record Dates: First submitted 2018-07-16; First posted 2018-08-02 (Actual); Last update posted 2018-08-02 (Actual); Status verified 2018-08

CONDITIONS: Xerostomia; Sjogren's Syndrome
Keywords: Xerostomia; Sjögren's syndrome; Topical dry mouth products; Olive Oil; Oral Health Impact Profile
MeSH Terms: conditions — Xerostomia; Sjogren's Syndrome

STUDY DESIGN:
Intervention Model Description: Randomized double-blind placebo controlled study
Who Masked: Participant, Care Provider
Masking Description: The study and placebo products had an identical appearance and were packaged identically. The sacs were numbered consecutively from 1 to 28. The company prepared and numbered the bag and all the participants were blinded to the treatment. Blinding was revealed after all participants finished the trial and all the data were collected.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test group (Experimental): Patients had to use:
  Mouthwash treatment (250 ml): Aqua, Betaine, Glycerin, PEG-40, Hydrogenated Castor Oil, Propylene Glycol, Xylitol, Aroma, Potassium Phosphate, Diazolidinyl Urea, Allantoin, Olea Europaea Fruit Oil, Sodium Methylparaben, Sodium Propylparaben, Sodium Fluoride, CI75810, Panthenol, Tocopheryl Acetate, Sucralose, Carum Petroselinum Seed Oil, Limonene.
  Toothpaste treatment (50 ml): Glycerin, Aqua, Hydrated Silica, Xylitol, Betine, Tetrapotassium Pyrophosphate, Olea Europaea Fruti Oil, Xanthan Gum, Titanium Dioxide, Potassium Phosphate, Aroma, Sodium Fluoride, Diazolidinyl Urea, Papain, Carum Petroselinum Seed Oil, Panthenol, Tocopheryl Acetate, Limonene
  Interventions: Other: Mouthwash treatment; Other: Toothpaste treatment
- Placebo group (Placebo Comparator): Patients had to use:
  Mouthwash placebo(250 ml): Aqua, Glycerin, PEG-40 Hydrogenated Castor Oil, Propylene Glycol, flavoring, Potassium Phospate, Diazolidinyl Urea, Sodium Methylparaben, Sodium Propylparaben, Sodium Fluoride, CI75810, Tocopheryl Acetate, Sucralose, LImonene.
  Toothpaste placebo (50 ml): Aqua, Sorbitol, Hydrated Silica, Glycerin, Tetrapotassium Pyrophosphate, Xanthan Gum Titanium Dioxide, Sodium Lauryl Sulphate, Potassium Phosphate, flavoring, Sodium Fluoride, Diazolidinyl Urea, Sucralose, Limonene
  Interventions: Other: Mouthwash placebo; Other: Toothpaste placebo

INTERVENTIONS:
Other: Mouthwash treatment — 60 seconds after meals (3 times/day) during 28 days
  Arms: Test group
Other: Toothpaste treatment — 3 minutes after the mouthwash (3 times/day) during 28 days
  Arms: Test group
Other: Mouthwash placebo — 60 seconds after meals (3 times/day) during 28 days
  Arms: Placebo group
Other: Toothpaste placebo — 3 minutes after the mouthwash (3 times/day) during 28 days
  Arms: Placebo group

SUMMARY:
Objectives: To assess the effects of topical dry mouth products (toothpaste and mouthwash) containing olive oil, parsley oil, provitamin B5, allantoin, betaine and xylitol in Primary Sjögren's syndrome patients with xerostomia.

Subjects and Methods: A double-blinded, placebo-controlled, randomized design where participants were randomly assigned at baseline test or placebo products. Participants used the products 3 times/day/28 days. The investigators used Visual Analog Scale for xerostomia and Oral Health Impact Profile-14, baseline and after treatment, to assess the possible improvement.

DETAILED DESCRIPTION:
The investigators conducted a randomized double-blind placebo controlled study among participants with Sjögren's syndrome who attended to the Oral Medicine Specialist Degree Program at the School of Dentistry at Complutense University in Madrid. The study was conducted in accordance to the principles of the Helsinki Declaration. This study followed the guidelines established by the Consort Statement.

Participants. All participants had a full medical history about Primary Sjögren's syndrome, where their rheumatologist detailed how the correct diagnosis was made according to American-European Consensus Group 2002 criteria. Demographic and Primary Sjögren's syndrome characteristics were collected. Stimulated and unstimulated whole saliva were collected following the drainage method at baseline by a single trained clinician blinded to the treatment. The saliva was collected before giving study instructions between 8-10 am. Hyposalivation was present when unstimulated whole saliva was less than 0.1 ml/min or stimulated whole saliva was less than 0.7 ml/min.

Preparations. The company Biocosmetics provided the test and placebo products. Placebo preparations were in identical white bottles (250mL) and white toothpastes (50mL) like study products. These preparations (study or placebo) did not contain irritant substances. The placebo included the same excipients resulting in solution similar to the experimental one in colour, flavour and density. All ingredients were equal in parts except the active products that were only present in the study products: betaine, xylitol, allantoin, Olea Europaea Fruit Oil (olive oil), Panthenol (provitamine B5) and Carum Petroselinum Seed oil (parsley oil). Test and placebo products contain sodium fluoride (mouthwash 250ppmF- and toothpaste 995ppmF-).

Interventions and instructions to participants. Participants were randomized to receive study or placebo mouthwash and toothpaste. Before starting treatment, participants were instructed to rinse with 7mL of mouthwash (study or placebo) for 60 seconds after meals (3 times/day). After rinsing the mouth, patients were instructed to brush their teeth with 0.5 g of study or placebo toothpaste following the Bass brushing technique for 3 minutes. We gave all the patients the same ultra soft dental brush (CS5460 Curaprox, Curaden AG, Kriens, Switzerland). The products had to be used for 28 days (4 weeks). Participants were informed that the use of any oral hygiene or xerostomia products apart from the intervention was prohibited. After giving the instructions, the investigators gave the patients the corresponding bag containing the study or placebo products, which was completely closed.

Sample size. The sample size was calculated considering a previous study that applied the same products. It was estimated that, at least, 50% of the test group would improve; so with an alpha of 0.05 and a statistical power of 80%, 12 subjects would be required in each group.

Randomisation. Participants were randomly assigned to one of treatments (study or placebo) in a 1:1 ratio using a computer-generated algorithm stratified by using a fixed block sized of 4. The company performed the randomisation and prepared the products in opaque bags following the results of randomization. The participants received the correspondence bag following the sequence of study entry.

Blinding. The study and placebo products had an identical appearance and were packaged identically. The sacs were numbered consecutively from 1 to 28. The company prepared and numbered the bag and all the participants were blinded to the treatment. Blinding was revealed after all participants finished the trial and all the data were collected.

Statistical methods. All the analysis was done using SPSS version 22.0 (SPSS Inc. New York, NY, USA). Statistical analysis included basic descriptive statistics. Comparison of continuous variables between test and placebo groups was done using Mann-Whitney U-test. Comparison of categorical variables was done using Chi-square test or Fisher's exact test. Wilcoxon signed-rank test was used to determine whether the intragroup decreases in Visual Analogue Scale and Oral Health Impact Profile 14 were statistically significant. Differences were considered significant if p was less than or equal to 0.05.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older, pSS patients diagnosed according to the AECG-2002 criteria, patients suffering xerostomia sensation, willingness to participate in the study, mentally and physical ability to participate and complete the study

Exclusion Criteria:

* patients who received or are being treated with head and neck radiotherapy, chemotherapy, pregnant and breast-feeding women and patients who were using other topical or systemic treatments for xerostomia.

Ages: 32 Years to 73 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2016-10-03 (Actual); Primary Completion 2017-11-02 (Actual); Study Completion 2017-11-30 (Actual)

PRIMARY OUTCOMES:
Changes in Validated visual analogue scale questionnaire for xerostomia | At baseline and day 28
  The questionnaire contained 8 items. Subjects marked a vertical line through a 10cm horizontal line to indicate their level of dryness in each question. The total score range from 0 to 80 cm.

SECONDARY OUTCOMES:
Changes in Oral patient's quality of life | At baseline and day 28
  The Spanish validated version of the Oral Health Impact Profile-14 questionnaire that included 14 questions about oral pain, physical, psychological, and social limitations and disabilities whose score range from 0 to 4 was used. The total score varies from 0 to 56. Poorer scores correspond to higher quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Rosa María López-Pintor, PhD, Study Director — Universidad Complutense Madrid

REFERENCES:
- [Background] Vitali C, Bombardieri S, Jonsson R, Moutsopoulos HM, Alexander EL, Carsons SE, Daniels TE, Fox PC, Fox RI, Kassan SS, Pillemer SR, Talal N, Weisman MH; European Study Group on Classification Criteria for Sjogren's Syndrome. Classification criteria for Sjogren's syndrome: a revised version of the European criteria proposed by the American-European Consensus Group. Ann Rheum Dis. 2002 Jun;61(6):554-8. doi: 10.1136/ard.61.6.554. PMID 12006334
- [Background] Navazesh M. Methods for collecting saliva. Ann N Y Acad Sci. 1993 Sep 20;694:72-7. doi: 10.1111/j.1749-6632.1993.tb18343.x. No abstract available. PMID 8215087
- [Background] Ship JA, McCutcheon JA, Spivakovsky S, Kerr AR. Safety and effectiveness of topical dry mouth products containing olive oil, betaine, and xylitol in reducing xerostomia for polypharmacy-induced dry mouth. J Oral Rehabil. 2007 Oct;34(10):724-32. doi: 10.1111/j.1365-2842.2006.01718.x. PMID 17824884
- [Background] Pai S, Ghezzi EM, Ship JA. Development of a Visual Analogue Scale questionnaire for subjective assessment of salivary dysfunction. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2001 Mar;91(3):311-6. doi: 10.1067/moe.2001.111551. PMID 11250628
- [Background] Montero-Martin J, Bravo-Perez M, Albaladejo-Martinez A, Hernandez-Martin LA, Rosel-Gallardo EM. Validation the Oral Health Impact Profile (OHIP-14sp) for adults in Spain. Med Oral Patol Oral Cir Bucal. 2009 Jan 1;14(1):E44-50. PMID 19114956